CLINICAL TRIAL: NCT00543959
Title: An Efficacy and Tolerability Study of MK0533 in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Brief Title: Efficacy and Tolerability of MK0533 in Patients With Type 2 Diabetes (0533-005)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study is being discontinued based on data suggesting that none of the doses tested demonstrated both glycemic & body fluid benefits vs. the comparitor
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0533-005; MK0533-005; 2007_544
Record Dates: First submitted 2007-10-05; First posted 2007-10-15 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- Part1 - Arm 1 (Experimental): Part1: Arm 1: drug
  Interventions: Drug: MK0533
- Part1 - Arm 2 (Placebo Comparator): Part1 - Arm 2: Pbo comparator
  Interventions: Drug: Comparator: Placebo (unspecified)
- Part 2 - Arm 1 (Placebo Comparator): Part 2 - Arm 1: Pbo
  Interventions: Drug: Comparator: Placebo (unspecified)
- Part 2 - Arm 2 (Experimental): Part 2- Arm 2: drug 5mg
  Interventions: Drug: MK0533
- Part 2 - Arm 3 (Experimental): Part 2 - Arm 3: drug 15mg
  Interventions: Drug: MK0533
- Part 2 - Arm 4 (Experimental): Part 2 - Arm 4: drug 30mg
  Interventions: Drug: MK0533
- Part 2 - Arm 5 (Active Comparator): Part 2 - Arm 5: active comparator
  Interventions: Drug: Comparator: pioglitazone

INTERVENTIONS:
Drug: MK0533 — Initially a 12-wk study of MK0533 30mg, switching at week 12 to a study of daily administration MK0533 5mg, MK0533 15mg, MK0533 30mg. Study period is a total of 24-wks.
  Arms: Part 2 - Arm 2; Part 2 - Arm 3; Part 2 - Arm 4; Part1 - Arm 1
Drug: Comparator: Placebo (unspecified) — MK0533 Placebo; MK0533 5mg; MK0533 15mg; MK0533 30mg. Study period is a total of 24 wks.
  Arms: Part 2 - Arm 1; Part1 - Arm 2
Drug: Comparator: pioglitazone — pioglitazone 45mg. Study period is a total of 24 wks.
  Arms: Part 2 - Arm 5

SUMMARY:
A study to evaluate the effectiveness and tolerability of MK0533 and pioglitazone in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 to 70 years with Type 2 diabetes who have not been able to adequately control their blood glucose levels
* Note: Only patients who have not been taking any antihyperglycemic medicine for 3 months will be screened

Exclusion Criteria:

* Patients taking any medicines that affect body fluid level such as a diuretic or water pill
* Patients taking niacin or other certain medications
* Patients with any of the following conditions: liver or kidney disease, poorly controlled high blood pressure, heart disease or certain blood disorders
* Patients with abnormal laboratory results from a blood test that will be given before each patient starts the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2006-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Body fluid gain from baseline after 12 weeks | 12 weeks

SECONDARY OUTCOMES:
Fasting plasma glucose after 12 weeks | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC